CLINICAL TRIAL: NCT02920788
Title: Multi-Level Assessment and Rehabilitation of Combat Mild TBI
Brief Title: Mild TBI Assessment & Rehabilitation
Acronym: MTAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N2300-R
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Brain Injuries, Traumatic
Keywords: Rehabilitation; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Therapeutics; Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Veteran Mild TBI Group - GOALS Intervention (Experimental): Veterans ages 18+ with chronic mild TBI, to undergo GOALS cognitive training as an intervention.
  Interventions: Behavioral: Goal-Oriented Attentional Self-Regulation (GOALS); Device: fMRI
- Veteran Mild TBI - Treatment as Usual (Active Comparator): Veterans ages 18+ with chronic mild TBI, matched by demographic and clinical criteria to the GOALS group, to receive the standard clinical care.
  Interventions: Other: Brain Health Education (BHE); Device: fMRI
- Veteran Non TBI - No Treatment (No Intervention): Veterans ages 18+ with no history of TBI, to undergo Neuropsychologic evaluation and MR Imaging with no intervention.

INTERVENTIONS:
Behavioral: Goal-Oriented Attentional Self-Regulation (GOALS) — GOALS is a manualized, therapist-administered cognitive training program that targets executive control functions of applied mindfulness-based attention regulation and goal management strategies and links them to participant-defined real-life goals. In contrast to training via practice on isolated tasks, this training protocol involves application of attention regulation skills and strategies to participant-defined goals in real life, ecologically valid settings. One of the main training aims is to improve self-regulatory control mechanisms as they contribute to goal attainment.
  Arms: Veteran Mild TBI Group - GOALS Intervention
Other: Brain Health Education (BHE) — BHE group is a formal in-person, active, psycho-educational, control intervention closely matched to GOALS for length, intensity, and contact with a therapist/facilitator. Topics include brain structure, function, sleep, stress, emotion and the brain.
  Other Names: Treatment As Usual (TAU)
  Arms: Veteran Mild TBI - Treatment as Usual
Device: fMRI — Functional Magnetic Resonance Imaging of the Brain
  Arms: Veteran Mild TBI - Treatment as Usual; Veteran Mild TBI Group - GOALS Intervention

SUMMARY:
One of the most pressing concerns within the VA currently is the provision of interventions that address the cognitive as well as emotional problems faced by Veterans with mild TBI and comorbid conditions. When completed, these studies will inform us whether training core attentional self-regulatory control functions via personally-relevant activities will be effective in improving daily life for Veterans with mild TBI and comorbid conditions. The study design will provide a test not only of potential benefits for real life functioning, but also determine to what extent these benefits are related to actual changes in cognitive/behavioral performance and brain networks corresponding to these functions. This project will provide a foundation for future studies to investigate the neural mechanisms that support improvements of cognition and behavior in mTBI.

DETAILED DESCRIPTION:
Combat-related mild traumatic brain injury (mTBI) and co-morbid conditions are prevalent in returning Veterans with the reported rates ranging from 14- 22%. Chronic sequela of mTBI can be highly debilitating due to deficits in the cognitive control processes, including attention, executive functions, and memory. In prior studies, individuals with chronic acquired brain injury who participated in a cognitive training program, Goal-Oriented Attentional Self-Regulation (GOALS), which targets executive control functions of applied mindfulness-based attention regulation and goal management, improved cognitive performance in areas of: complex attention/executive function and memory, complex functional task performance, and daily functioning. Furthermore, functional MRI (fMRI) results after training indicated significantly enhanced modulation of neural processing. Preliminary data from recently completed randomized-control GOALS study in 32 Veterans with chronic TBI also show both short and longer term (up to 2 years) improvements in attention and executive function, complex real-life tasks, and emotional regulation.

The primary objectives of this study are to investigate the potential short and longer term effects of GOALS cognitive training program, and to use advanced MRI to investigate changes in brain structure and function in the circuits that regulate attention, memory, executive function and emotion in Veterans with chronic mTBI.

The investigators postulate that 1) GOALS training will improve neurocognitive function in attention and executive function domains, complex functional task performance, and emotional regulation in Veterans with chronic mTBI; 2) improved neurocognitive function will be correlated with macrostructural, microstructural and functional changes in the corresponding brain networks on high field (3T) and ultra-high field (7T) structural MR imaging, diffusion tensor imaging (DTI) and resting state fMRI performed pre- and post-training; 3) Changes in both behavioral function and imaging measures will be maintained at 6 months post-training and be associated with improvements in activities and participation.

AIM 1: To determine the short and long term effects of GOALS training on neuro-cognitive performance and neural plasticity of attention and executive control networks in mTBI.

AIM 2: To determine the short and long term effects of GOALS training on complex functional task performance and daily functioning, and on plasticity in pathways related to memory function, in mTBI.

AIM 3: To determine the short and long term effects of GOALS training on measures of emotional regulation, and on plasticity of frontolimbic networks related to emotion processing, in mTBI In a randomized, controlled interventional study design, 36 Veterans with a history of chronic (> 6 month) mTBI and residual cognitive difficulties will be randomized to participate in 5 weeks of cognitive training (GOALS) or a treatment as usual (TAU) comparison. At baseline, week 5 (post GOALS), and at 6 months, participants will undergo a multi-level assessment battery consisting of: 1) neuroimaging with high field (3T) and ultra-high field (7T) structural MR imaging, diffusion tensor imaging (DTI) and resting state fMRI; 2) neuropsychological assessment focusing on complex attention and executive function; 3) complex 'real life' functional task performance; and 4) self-report measures of daily functioning and emotional regulation/health.

Additionally, the investigators will be recruiting a separate cohort of 15 equally matched healthy veteran volunteers who have no TBI history, for normative comparisons. TBI-negative participants, who will not be participating in training sessions, will have neuroimaging with ultra-high field (7T) structural MR imaging and neuropsychological assessments at baseline and week 5.

When completed, this project will determine whether training core attentional self-regulatory control functions via personally-relevant activities will be effective in improving quality of life and daily functioning for Veterans with mTBI. The study design will provide a test of potential benefits on real-life functioning, and also determine to what extent these benefits are related to actual changes in hypothetically targeted cognitive/behavioral functions and brain networks corresponding to these functions.

Overall recruitment status was changed due to a new study site being added at UCSF. This was made possible by funding recently received from private donation through UCSF's Weill Institute for Neuroscience to study a cohort recruited via physician referral at UCSF.

ELIGIBILITY:
Inclusion Criteria:

For TBI-positive veteran participants, to be randomized to either GOALS or TAU:

* Ages 18+
* A history of mild TBI (as defined by DOD / VA; confirmed by medical records and in person Ohio State University TBI Instrument)
* Chronic, stable phase of recovery (>6 months from last post-concussive event)
* Report of residual cognitive difficulties (1 moderate or severe cognitive symptom(s) on the Neurobehavioral Symptom Inventory (NSI)) that interfere(s) with daily function
* Able and willing to commit to participate in training and assessments
* If on psychoactive medications, must be stable on medications (> 30 days)

For the TBI-negative healthy veteran control group:

* Ages 18+
* No history of any (mild to severe) TBI (as defined by DOD / VA; confirmed by medical records and in person Ohio State University TBI Instrument)
* Able and willing to commit to participate in assessments
* If on psychoactive medications, must be stable on medications (> 30 days)

Exclusion Criteria:

For the TBI-positive veteran participants, to be randomized to either GOALS or TAU:

* A history of moderate or severe TBI
* Unstable medical, neurologic, or psychiatric condition, including severe cognitive dysfunction, or other reasons for being unable or unwilling to participate in study procedures (e.g., contraindications to MRI)
* Ongoing illicit drug or alcohol abuse (AUDIT>8)
* Psychosis
* Severe depression, anxiety or PTSD that precludes participation in research activities
* Poor English comprehension
* Eligible participants may have other co-morbid stable neuropsychiatric disorders, including depression and PTSD
* There will be no restriction in regard to gender, race and socioeconomic status

For the TBI-negative healthy veteran control group:

* A history of any mild, moderate, or severe TBI
* Unstable medical, neurologic, or psychiatric condition, including severe cognitive dysfunction, or other reasons for being unable or unwilling to participate in study procedures (e.g. contraindications to MRI)
* Ongoing illicit drug or alcohol abuse (AUDIT>8)
* Psychosis
* Severe depression, anxiety or PTSD that precludes participation in research activities
* Poor English comprehension
* Eligible participants may have other co-morbid stable neuropsychiatric disorders, including depression and PTSD.
* There will be no restriction in regard to gender, race and socioeconomic status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Delis-Kaplan Executive Function System (D-KEFS) Stroop Inhibition-Switching Task | 6 months after enrollment
  Single Test for Attention, Executive Function and Mental Flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Pratik Mukherjee, MD PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Novakovic-Agopian T, Kornblith E, Abrams G, Burciaga-Rosales J, Loya F, D'Esposito M, Chen AJW. Training in Goal-Oriented Attention Self-Regulation Improves Executive Functioning in Veterans with Chronic Traumatic Brain Injury. J Neurotrauma. 2018 Dec 1;35(23):2784-2795. doi: 10.1089/neu.2017.5529. Epub 2018 Jul 23. PMID 29717652
- [Result] Kryza-Lacombe M, Santiago R, Hwang A, Raptentsetsang S, Maruyama BA, Chen J, Cassar M, Abrams G, Novakovic-Agopian T, Mukherjee P. Resting-State Connectivity Changes After Goal-Oriented Attentional Self-Regulation Training in Veterans With Mild Traumatic Brain Injury: Preliminary Findings from a Randomized Controlled Trial. Neurotrauma Rep. 2023 Jun 29;4(1):420-432. doi: 10.1089/neur.2022.0074. eCollection 2023. PMID 37405257
- [Result] Karbasforoushan H, Wren-Jarvis J, Hwang A, Santiago R, Raptentsetsang S, Cai LT, Xiao J, Maruyama BA, Abrams GM, Novakovic-Agopian T, Mukherjee P. Goal-Oriented Attentional Self-Regulation Training in Chronic Mild Traumatic Brain Injury is Linked to Microstructural Plasticity in Prefrontal White Matter. J Neurotrauma. 2025 Jan;42(1-2):46-56. doi: 10.1089/neu.2023.0229. Epub 2024 Oct 29. PMID 39470361
- [Result] Novakovic-Agopian T, Posecion L, Kornblith E, Abrams G, McQuaid JR, Neylan TC, Burciaga J, Joseph J, Carlin G, Groberio J, Maruyama B, Chen AJW. Goal-Oriented Attention Self-Regulation Training Improves Executive Functioning in Veterans with Post-Traumatic Stress Disorder and Mild Traumatic Brain Injury. J Neurotrauma. 2021 Mar;38(5):582-592. doi: 10.1089/neu.2019.6806. Epub 2020 Nov 18. PMID 33019861